CLINICAL TRIAL: NCT07010094
Title: A Prospective, Multicenter, Single-arm, Target-Value Clinical Trial to Evaluate the Safety and Efficacy of BM Shockwave Devices to Treat Coronary Calcified Lesions
Brief Title: BM Shockwave Devices Clinical Study in Coronary Calcified Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D24
Record Dates: First submitted 2025-05-28; First posted 2025-06-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; shockwave therapy; Coronary calcified lesions
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental)
  Interventions: Device: BM shockwave devices

INTERVENTIONS:
Device: BM shockwave devices — Use the BM shockwave devices for pre-treatment of coronary calcification lesions.

SUMMARY:
This clinical trial is a prospective, multicenter, single-arm, target-value study to verify the safety and efficacy of BM coronary shockwave devices for the treatment of coronary calcification lesions.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  1. Age 18-85 years, male or female;
  2. Patients with evidence of asymptomatic ischemia, stable or unstable angina, or old myocardial infarction;
  3. Patient is able and willing to comply with all assessments in the study.

Angiography inclusion criteria:

1. The target lesion is a de novo, in-situ coronary artery lesion;
2. The target lesion length is ≤40 mm, and the target lesion reference vessel diameter is 2.0-4.0 mm (visual estimation);
3. The target lesion diameter stenosis is visually estimated to be ≥70%, or <70% but ≥50% with evidence of ischemia;
4. Clear high-density calcification shadows are visible both during cardiac contraction and at rest;
5. Target vessel TIMI flow grade 3 prior to use of the investigational device (pre-dilatation is permitted);
6. The target lesion is the only calcified lesion to be treated with shock wave therapy in this session; if non-target lesions are present, they must be successfully treated prior to the target lesion;
7. Patients suitable for treatment with metal stent implantation.

Exclusion Criteria:

* General exclusion criteria:

  1. ST-segment elevation myocardial infarction within 3 days prior to the procedure;
  2. Use of rotational atherectomy or special balloons (chocolate balloon, scoring balloon, cutting balloon, etc.) for lesion pretreatment;
  3. New York Heart Association (NYHA) functional class III or IV;
  4. Target lesion expected to require full biodegradable scaffold implantation, drug-eluting balloon dilation, or percutaneous transluminal coronary angioplasty (PTCA) treatment;
  5. Uncontrolled severe hypertension (persistent: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg);
  6. Severe liver or kidney dysfunction, with transaminase levels exceeding three times the upper limit of normal, serum creatinine >2.5 mg/dL (221 μmol/L), or chronic kidney failure requiring long-term dialysis;
  7. Platelet count <60 × 10⁹/L;
  8. Stroke within the past 6 months prior to enrollment, excluding transient ischemic attack (TIA) and lacunar infarction;
  9. Active peptic ulcer or history of upper gastrointestinal bleeding within the past 6 months prior to enrollment;
  10. Known allergy to heparin, contrast agents, aspirin, clopidogrel, or anesthetics;
  11. Patients with a life expectancy of less than 12 months due to severe medical conditions;
  12. Patients who have participated in other drug or device clinical trials and failed to meet the primary endpoint;
  13. Pregnant or breastfeeding women;
  14. Patients deemed by the investigator to have poor compliance and unable to complete the study according to the protocol.

Contrast exclusion criteria:

1. The target lesion and non-target lesion are in the same vascular branch;
2. The target lesion is at the origin (LAD, LCX, or RCA, within 5 mm of the origin) or an unprotected left main lesion;
3. A stent has been implanted within 10 mm of the proximal or distal end of the target lesion;
4. The target lesion has an unprotected branch vessel with a diameter of 2.5 mm or greater;
5. The target lesion is located distal to the saphenous vein or LIMA (left internal mammary artery)/RIMA (right internal mammary artery) bypass graft;
6. An aneurysm is present within 10 mm of the target lesion;
7. Contrast imaging confirms the presence of an NHLBI classification D-F type arterial dissection at the target lesion prior to the use of the investigational device;
8. The target lesion has definite thrombus formation;
9. The investigator determines that the target lesion is not suitable for vascular dilation in the patient.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure success rate | Endpoints will be measured through hospital discharge (expected to be within 7 days)
  Definition: Residual stenosis ≤30% after PCI, and no major adverse cardiac events (MACE) events occurring during hospitalization. MACE is defined as cardiac death, myocardial infarction, and target vessel revascularization events.

SECONDARY OUTCOMES:
Angiography success rate | 0 day
  Definition: After successful stent placement in the target lesion, residual stenosis ≤ 30%, and no serious angiography complications occur.
  Serious angiography complications: refer to the occurrence of D-F type dissection, vascular perforation, acute vascular occlusion, persistent slow blood flow, or no reperfusion during the procedure.
Device success rate | 0 day
  The study device successfully passes through the target lesion, and no serious angiographic complications occur immediately after shockwave pretreatment.
Residual stenosis | 0 day
  Degree of residual stenosis immediately after shockwave pretreatment of the target lesion.
MACE rate | 30 days
  MACE is defined as cardiac death, myocardial infarction, and target vessel revascularization events.
Target lesion failure | 30 days
  Target lesion failure (TLF) definition: Includes cardiac death, myocardial infarction caused by target vessel (ST-segment elevation or non-ST-segment elevation myocardial infarction), and target lesion revascularization.
Device defects | 0 day
  Incidence of device defects

CONTACTS AND LOCATIONS:
Locations (1):
- Xiamen University Affiliated Cardiovascular Hospital, Fujian, Xiamen, China

IPD SHARING:
Plan to Share IPD: No